CLINICAL TRIAL: NCT03226106
Title: Optimizing Physical Activity Outcomes for Veterans After Total Knee Arthroplasty
Brief Title: Optimizing Physical Activity Outcomes After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F2417-R
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Total Knee Arthroplasty; Osteoarthritis
Keywords: Rehabilitation; Total Knee Arthroplasty; Telemedicine; Physical Activity
MeSH Terms: conditions — Osteoarthritis; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial; Two groups.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical Activity Behavior Intervention (Experimental): A 12-week behavior change intervention that supplements conventional rehabilitation including: 10 telerehabilitation sessions, daily activity sensor use, education, self-monitoring, tailored feedback, barrier/facilitator identification, promotion of problem solving, action planning, and encouragement.
  Interventions: Behavioral: Physical Activity Behavior Intervention
- Attention Control (Active Comparator): Conventional rehabilitation with 10 telerehabilitation sessions that match the frequency and duration of the experimental arm. Attention control intervention provided as 10 telerehabilitation sessions of non-physical activity related education-only sessions.
  Interventions: Other: Attention Control

INTERVENTIONS:
Behavioral: Physical Activity Behavior Intervention — Home-based weekly sessions (30 min) using behavior change methods for promoting physical activity. Sessions will occur using home-based computer tablets for real-time video interface between the participant and researcher. Participants will wear wrist-mounted activity sensors with direct physical activity feedback during the intervention period to allow for behavioral feedback and action planning.
  Arms: Physical Activity Behavior Intervention
Other: Attention Control — Conventional rehabilitation with supplemental 10 telerehabilitation sessions that match the frequency and duration of the experimental arm. Attention control intervention provided as 10 telerehabilitation sessions of non-physical activity related education-only sessions.
  Arms: Attention Control

SUMMARY:
Although total knee arthroplasty is an effective intervention for decreasing knee pain and improving physical function, physical activity levels remain low up to a year after surgery. This study will use mobile-health technology to deliver an intervention designed to improve physical activity behavior for Veterans recovering from total knee arthroplasty. The study will assess the effectiveness of using behavior-change intervention as a supplement to conventional rehabilitation to improve physical activity. The intervention will be delivered using home-based tablet computers for Veterans to have remote interaction with the researcher and real-time physical activity feedback from a wrist-worn activity sensor.

DETAILED DESCRIPTION:
This randomized clinical trial will assess the efficacy of using physical activity behavior change intervention for Veterans recovering from total knee arthroplasty. Testing will occur at baseline (before surgery), at intervention midpoint (8 weeks after surgery), end of intervention (14 weeks after surgery), and 24 weeks after intervention. The primary outcome is accelerometer-assessed daily step count. Secondary outcomes include the percent time engaged in standing and walking activity and physical function (Six-Minute Walk, 30-Second Chair-Stand Test, Timed Up-and-Go, Western Ontario and McMaster Universities Osteoarthritis Index, and the Veterans RAND 12-Item Health Survey.

ELIGIBILITY:
Inclusion Criteria:

* Veteran
* Planned unilateral total knee arthroplasty

Exclusion Criteria:

* Severe non-surgical limb pain (pain >5/10 on non-surgical limb with walking)
* Unstable orthopedic, neurologic, or pulmonary condition that limits function
* Unstable cardiac condition
* Uncontrolled hypertension
* Uncontrolled diabetes
* Acute systemic infection
* Active cancer treatment
* Recent stroke (within 2 years)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cory L. Christiansen, PhD, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (1):
- Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be made available at time of study completion, per VA recommendations and approval.

REFERENCES:
- [Background] Kline PW, Melanson EL, Sullivan WJ, Blatchford PJ, Miller MJ, Stevens-Lapsley JE, Christiansen CL. Improving Physical Activity Through Adjunct Telerehabilitation Following Total Knee Arthroplasty: Randomized Controlled Trial Protocol. Phys Ther. 2019 Jan 1;99(1):37-45. doi: 10.1093/ptj/pzy119. PMID 30329126
- [Background] Hoffman RM, Davis-Wilson HC, Hanlon S, Swink LA, Kline PW, Juarez-Colunga E, Melanson EL, Christiansen CL. Maximal daily stepping cadence partially explains functional capacity of individuals with end-stage knee osteoarthritis. PM R. 2024 Jun;16(6):532-542. doi: 10.1002/pmrj.13082. Epub 2023 Nov 27. PMID 37819260

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 114 participants were enrolled in the study. There were n=22 participants lost to follow-up before randomization: n=14 post-consent screen fail, n=7 withdrew, and n=1 no valid baseline activity data. n=92 participants were randomized in the study.
Period: Overall Study
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Started | 46 | 46
Week 8 | 43 | 46
Week 14 (Intervention End) | 43 | 46
Completed | 41 | 46
Not Completed | 5 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: US military Veterans (aged 50-85 years) scheduled for unilateral TKA.
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Behavior Intervention | Attention Control | Total
Number analyzed (Participants) | 46 | 46 | 92
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [63 to 72] | 68 [60 to 71] | 68 [62 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 3 | 11
  Male | 38 | 43 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 12 | 18
  Not Hispanic or Latino | 36 | 32 | 68
  Unknown or Not Reported | 4 | 2 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 7 | 4 | 11
  Caucasian | 38 | 39 | 77
  Other | 0 | 2 | 2
  Unknown or Not Reported | 1 | 1 | 2
Education [Count of Participants; unit: Participants]
  < High School / High School | 15 | 20 | 35
  Bachelor or Associate Degree | 22 | 21 | 43
  Master's or Professional Degree | 7 | 4 | 11
  Other | 1 | 1 | 2
  Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Free-living Daily Step Count
Description: Accelerometer-based measurement of free-living daily step count
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: step count
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
step count | 6947 [4656 to 8825] | 6339 [4851 to 8145]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.024, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; We used a linear mixed model with a random intercept for subject and fixed effects for age, time, and interaction between intervention arm and time; Mean Difference (Final Values) = 930.51, 95% CI 2-sided [41.65 to 1819.36] — The difference is the estimated mean between the intervention and control arms

2. Secondary Outcome: 30-Second Chair-Stand Test W14
Description: Physical function test that assesses the number of sit-stand-sit transitions that a participant performs in the span of 30 seconds.
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: sit-stand-sit transitions
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
sit-stand-sit transitions | 13 [10 to 14] | 12 [9 to 15]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.584, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.70, 95% CI 2-sided [-0.67 to 2.07] — The difference is the estimated mean between the intervention and control arms

3. Secondary Outcome: 30-Second Chair-Stand Test W38
Description: as for outcome 2
Time Frame: 24 weeks after intervention (week 38 of study)
Measure: Mean (Inter-Quartile Range); unit: sit-stand-sit transitions
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
sit-stand-sit transitions | 14 [12 to 16] | 14 [11 to 16]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.724, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-1.40 to 1.32] — The difference is the estimated mean between the intervention and control arms

4. Secondary Outcome: Six-Minute Walk Test W14
Description: Physical function test measuring the total distance walked in a span of six minutes.
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: meters
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
meters | 433 [391 to 478] | 434 [365 to 515]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.547, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.49, 95% CI 2-sided [-18.90 to 33.89] — The difference is the estimated mean between the intervention and control arms

5. Secondary Outcome: Six-Minute Walk Test W38
Description: Physical function test measuring the total distance walked in a span of six minutes.
Time Frame: 24 weeks after intervention (week 38 of study)
Measure: Mean (Inter-Quartile Range); unit: meters
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
meters | 452 [427 to 488] | 451 [379 to 489]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.716, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.93, 95% CI 2-sided [-21.67 to 31.54] — The difference is the estimated mean between the intervention and control arms

6. Secondary Outcome: Timed Up-and-Go Test W14
Description: A physical performance measure that includes rising from a chair, walking 3 meters, turning 180 degrees, returning to chair, and sitting.
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
seconds | 9.8 [8.2 to 9.7] | 9.4 [7.8 to 10.9]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.946, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.88 to 0.82] — The difference is the estimated mean between the intervention and control arms

7. Secondary Outcome: Timed Up-and-Go Test W38
Description: as for outcome 6
Time Frame: 24 weeks after intervention (week 38 of study)
Measure: Mean (Inter-Quartile Range); unit: seconds
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
seconds | 9.1 [7.4 to 9.7] | 9.0 [7.5 to 10.3]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.906, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-1.08 to 0.52] — The difference is the estimated mean between the intervention and control arms

8. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index W14
Description: Self-report health status measure of pain, stiffness, and function for people with osteoarthritis of the hip or knee. A higher score indicates worse outcome with the Total Score range from 0-96. A positive change indicates worse outcome and a negative change indicates a better outcome across time points.
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
score on a scale | 18 [5 to 26] | 21 [12 to 30]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.873, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.55, 95% CI 2-sided [-7.59 to 4.49] — The difference is the estimated mean between the intervention and control arms

9. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index W38
Description: as for outcome 8
Time Frame: 24 weeks after intervention (week 38 of the study)
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
score on a scale | 13 [2 to 22] | 22 [6 to 34]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.241, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.26, 95% CI 2-sided [-12.48 to -0.04] — The difference is the estimated mean between the intervention and control arms

10. Secondary Outcome: Veterans RAND 12-Item Health Survey Physical Component W14
Description: A self-report assessment of health-related quality of life assessing the domains of physical functioning, role-physical, bodily pain, general health perceptions, vitality, social functioning, role-emotional, and mental health. All items are scored so that a high score defines a more favorable health state. In addition, each item is scored on a 0 to 100 range so that the lowest and highest possible scores are 0 and 100, respectively. Scores represent the percentage of total possible score achieved.
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: Percentage of total
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
Percentage of total | 43 [38 to 50] | 39 [34 to 45]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.223, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.86, 95% CI 2-sided [-0.39 to 6.12] — The difference is the estimated mean between the intervention and control arms

11. Secondary Outcome: Veterans RAND 12-Item Health Survey Physical Component W38
Description: as for outcome 10
Time Frame: 24 weeks after intervention (week 38 of study)
Measure: Mean (Inter-Quartile Range); unit: Percentage of total
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
Percentage of total | 43 [39 to 52] | 41 [35 to 49]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.388, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.17, 95% CI 2-sided [-2.19 to 4.53] — The difference is the estimated mean between the intervention and control arms

12. Secondary Outcome: Veterans RAND 12-Item Health Survey Mental Component W14
Description: as for outcome 10
Time Frame: End of intervention (14 weeks)
Measure: Mean (Inter-Quartile Range); unit: Percentage of total
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 43 | 46
Percentage of total | 54 [48 to 60] | 52 [44 to 60]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.88, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-4.08 to 2.68] — The difference is the estimated mean between the intervention and control arms

13. Secondary Outcome: Veterans RAND 12-Item Health Survey Mental Component W38
Description: as for outcome 10
Time Frame: 24 weeks after intervention (week 38 of study)
Measure: Mean (Inter-Quartile Range); unit: Percentage of total
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
Percentage of total | 55 [52 to 59] | 51 [42 to 60]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.85, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.77, 95% CI 2-sided [-2.63 to 4.17] — The difference is the estimated mean between the intervention and control arms

14. Secondary Outcome: Free-living Daily Step Count W38
Description: Accelerometer-based measurement of free-living daily step count
Time Frame: 24 weeks after intervention (week 38 of study)
Measure: Mean (Inter-Quartile Range); unit: step count
Arm/Group | Physical Activity Behavior Intervention | Attention Control
Number analyzed (Participants) | 41 | 46
step count | 7287 [4279 to 9630] | 6855 [4441 to 9118]
Statistical Analysis 1: Comparison: Physical Activity Behavior Intervention vs Attention Control; Test type: Superiority; p = 0.101, Mixed Models Analysis — The value corresponds to the interaction between time and group assignment; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 559.81, 95% CI 2-sided [-405.01 to 1524.62] — The difference is the estimated mean between the intervention and control arms

ADVERSE EVENTS:
Time Frame: Adverse events were collected between baseline testing (pre-surgery) through the end of the study at 38 weeks post-surgery.
Description: Adverse events were collected throughout the study and categorized using the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Arm/Group | Physical Activity Behavior Intervention | Attention Control
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/46
Serious Adverse Events (participants affected / at risk) | 3/46 | 8/46
Other Adverse Events (participants affected / at risk) | 33/46 | 43/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Behavior Intervention (N=46) | Attention Control (N=46)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gastrointestinal Disorders (Gastrointestinal disorders) | 0 (0) | 1 (1)
General disorders and administration site conditions (General disorders) | 1 (1) | 0 (0)
Musculoskeletal & connective tissue disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous System Disorders (Nervous system disorders) | 1 (1) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Physical Activity Behavior Intervention (N=46) | Attention Control (N=46)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 11 (22) | 15 (28)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorders (Cardiac disorders) | 1 (1) | 0 (0)
Eye disorders (Eye disorders) | 1 (1) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 2 (2) | 2 (2)
General disorders and administration site conditions (General disorders) | 4 (4) | 5 (7)
Immune system disorders (Immune system disorders) | 1 (1) | 0 (0)
Infections and infestations (Infections and infestations) | 2 (2) | 4 (4)
Musculoskeletal & connective tissue disorders (Musculoskeletal and connective tissue disorders) | 5 (6) | 8 (11)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 0 (0) | 1 (1)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 2 (2)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
Vascular disorder (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-18): https://cdn.clinicaltrials.gov/large-docs/06/NCT03226106/Prot_SAP_001.pdf
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT03226106/ICF_000.pdf